CLINICAL TRIAL: NCT01323309
Title: A Randomized Controlled Trial of Individual Psychosocial Interventions for Cancer Patients
Brief Title: Trial of Individual Psychosocial Interventions for Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fordham University (Other)
Responsible Party: Sponsor
Other Study IDs: 11-021
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor Diseases
Keywords: Supportive Psychotherapy; Therapy; 11-021

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Individual Meaning-Centered Psychotherapy (IMCP)
  Interventions: Behavioral: Individual Meaning-Centered Psychotherapy (IMCP)
- standard Individual Supportive Psychotherapy (ISP)
  Interventions: Behavioral: standard Individual Supportive Psychotherapy (ISP)
- enhanced usual care (EUC)
  Interventions: Behavioral: enhanced usual care (EUC)

INTERVENTIONS:
Behavioral: Individual Meaning-Centered Psychotherapy (IMCP) — IMCP is based on the principles of Viktor Frankl's Logotherapy, and is designed to help patients with advanced cancer sustain or enhance a sense of meaning, peace and purpose in their lives even as they approach the end of life. IMCP is structured as a 7-session (1-hour weekly sessions) individual intervention that utilizes a mixture of didactics, discussion and experiential exercises that focus around particular themes related to meaning and advanced cancer. In addition we will be asking patients in the IMCP arm to complete an optional weekly session rating survey
  Groups: Individual Meaning-Centered Psychotherapy (IMCP)
Behavioral: standard Individual Supportive Psychotherapy (ISP) — The ISP intervention utilized as the comparison treatment condition in this study, is adapted from the Supportive Group Psychotherapy manualized intervention developed by David Payne (1997) and adapted by Drs. Kissane, Breitbart and colleagues into the ISP manualized intervention. This intervention is a 7-session individual supportive psychotherapy utilizing an approach to supportive psychotherapy based on models described by Rogers. The essential components of supportive psychotherapy are integrated into this manualized intervention, including: reassurance, explanation, guidance, suggestion, encouragement, affecting changes in patient's environment, and permission for catharsis.
  Groups: standard Individual Supportive Psychotherapy (ISP)
Behavioral: enhanced usual care (EUC) — We are therefore including what we refer to as an "enhanced" usual care arm to this randomized controlled trial to address the ethical issues raised by utilizing a usual care condition in a vulnerable advanced cancer population. Participants will receive feedback about their level of distress (based on the DT administered at screening) and given appropriate targeted referrals based on levels of distress and problem areas endorsed. Participants will be given a letter with a list of appropriate referrals.
  Other Names: Several referrals may be made based on identified problem areas, using the following guidelines:; • "Practical Problems" - Social Work on their disease management team; • "Family Problems"- Family Clinic at MSKCC Counseling Center; • "Emotional Problems" - MSKCC Counseling Center; • "Spiritual/Religious Concern"- Pastoral Care Counseling Services; • "Physical Problems"- MSKCC physician or MSKCC Palliative Care Service
  Groups: enhanced usual care (EUC)

SUMMARY:
The aim of the study is to compare the benefits of three types of individual treatment programs for cancer patients: Meaning-Centered counseling, Supportive counseling, and Enhanced Usual Care.

We would like to train therapists in administering these types of counseling, so that they have expertise to work on the study. The therapists will administer either the Meaning-Centered counseling or the Supportive counseling, as part of their training.

Many cancer patients use counseling or other resources to help with the emotional burden of their illnesses. Counseling often helps them cope with cancer by giving them a place to express their feelings. "Meaning-Centered" counseling aims to teach cancer patients how to maintain or even increase a sense of meaning and purpose in their lives, despite cancer. "Supportive" counseling is intended to help the patient cope with cancer by giving them a place to express their feelings and get support. Enhanced Usual Care is intended to offer the patient referrals and resources that are matched to their individual needs in addition to the care they are already receiving at MSKCC.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* Able to communicate and understand English well enough to complete assessments and intervention**
* Patients solid tumors with advanced disease receiving ambulatory care at MSKCC*.
* Distress Thermometer rating of 4 or greater*

  * Patients who do not meet these eligibility criteria may be offered participation as a training case (See inclusion criteria for Training Cases below).

Subject Inclusion Criteria- Training Cases

* 21 years of age and older
* Able to communicate and understand English well enough to complete the intervention**
* Patients with solid tumors with advanced disease receiving ambulatory care at MSKCC with a Distress Thermometer rating of 3 or less. or Patients with solid tumors who do not meet eligibility criteria for advanced disease receiving ambulatory care at MSKCC.

or Patients solid tumors with advanced disease receiving ambulatory care at MSKCC who have participated in a prior meaning focused intervention study. or Patients with solid tumors with advanced disease receiving ambulatory care at MSKCC who have enrolled in this study, been assigned to the EUC arm, and completed all study requirements including follow-up assessments.

**The study treatment manual materials and assessments were designed and validated in English and are not currently available in other languages. Translation of the intervention and questionnaires into other languages would require reestablishing the reliability and validity of them. Therefore, participants must be able to communicate in English.

Exclusion Criteria:

* In the judgment of the treating physician and/or the consenting professional, presence of significant cognitive impairment (i.e., delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection.
* Baseline Karnofsky Performance Rating Scale (KPRS) score below 60 or physical limitations sufficient to preclude participation in a 7 session outpatient psychotherapy intervention.
* In the judgment of the consenting professional, severe psychiatric disturbance sufficient that would preclude participation in the intervention (patients whose psychiatric disorder is well controlled on medication will be eligible).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential candidates for the study who meet the eligibility criteria of cancer diagnosis and stage will be identified by the research staff and/or participating oncology staff or co-investigators. Study investigators in the Pain & Palliative Care Service the Breast Cancer Medicine Service, the Head & Neck Oncology Service, the Thoracic Medicine Service, the Gastrointestinal Oncology Service, and the Genito-Urinary Oncology Service will serve as liaisons to the Research Staff and help screen and identify potential subjects for the study.
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2011-03-22 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Marziliano A, Applebaum A, Moyer A, Pessin H, Rosenfeld B, Breitbart W. The Impact of Matching to Psychotherapy Preference on Engagement in a Randomized Controlled Trial for Patients With Advanced Cancer. Front Psychol. 2021 Feb 24;12:637519. doi: 10.3389/fpsyg.2021.637519. eCollection 2021. PMID 33732196
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individual Meaning-Centered Psychotherapy (IMCP) | Standard Individual Supportive Psychotherapy (ISP) | Enhanced Usual Care (EUC)
Started | 109 | 108 | 104
Completed | 70 | 54 | 53
Not Completed | 39 | 54 | 51
Not completed — Death | 9 | 15 | 5
Not completed — Lost to Follow-up | 11 | 14 | 24
Not completed — Withdrawal by Subject | 14 | 14 | 18
Not completed — Disease progression | 5 | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Meaning-Centered Psychotherapy (IMCP) | Standard Individual Supportive Psychotherapy (ISP) | Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 109 | 108 | 104 | 321
Age, Continuous [Mean (Full Range); unit: years] | 58.1 [33 to 84] | 58.8 [25 to 83] | 57.1 [25 to 85] | 58.0 [25 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 71 | 78 | 230
  Male | 28 | 37 | 26 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 14 | 30
  Not Hispanic or Latino | 100 | 100 | 89 | 289
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 11 | 7 | 33
  White | 87 | 85 | 88 | 260
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 8 | 5 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109 | 108 | 104 | 321

OUTCOME MEASURES:

1. Primary Outcome: Participant Meaning Making Scores Using the Life Attitude Profile-Revised (LAP-R)
Description: The Life Attitude Profile-Revised (LAP-R) is a 48-item self-report measure of discovered meaning and purpose in life and the motivation to find meaning and purpose in life. There are 6 subscales: Purpose (8 items, Minimum 8, Maximum 56, Higher is better), Coherence (8 items, Minimum 8, Maximum 56, Higher is better), Life control (8 items, Minimum 8, Maximum 56, Higher is better), Death acceptance (8 items, Minimum 8, Maximum 56, Higher is better), Existential transcendence (16 items, Minimum 16, Maximum 112, Higher is better), Personal Meaning (16 items, Minimum 16, Maximum 112, Higher is better), Goal Seeking (8 items, Minimum 8, Maximum 56, Higher is better): LAP-R total score (48 items, Minimum 72, Maximum 504, Higher is better). The LAP-R total score is derived by summing all subscales.
Time Frame: baseline meaning making measures and again at post-intervention (approximately week 8)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Individual Meaning-Centered Psychotherapy (IMCP) | Standard Individual Supportive Psychotherapy (ISP) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 94 | 86 | 74
scores on a scale
  Purpose at Baseline | 37.07 (9.33) | 38.28 (8.25) | 36.80 (9.11)
  Purpose at Post-intervention | 42.22 (8.77) | 41.09 (7.70) | 37.40 (7.78)
  Coherence at Baseline | 37.67 (9.97) | 38.73 (9.14) | 38.69 (8.29)
  Coherence at Post-intervention | 43.60 (8.86) | 41.39 (8.19) | 40.55 (8.60)
  Personal meaning at Baseline | 74.74 (18.03) | 77.01 (15.95) | 75.49 (16.26)
  Personal meaning at Post-intervention | 85.82 (16.84) | 92.48 (14.72) | 77.95 (14.96)
  Existential Transcendence at Baseline | 78.27 (33.14) | 79.42 (32.99) | 75.66 (30.26)
  Existential Transcendence at Post-intervention | 102.27 (33.14) | 91.07 (31.24) | 80.97 (30.80)

2. Secondary Outcome: Clinical and Demographic Variables That May Correspond to Differential Responses to Individual Meaning-Centered Psychotherapy
Description: The Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Scale (SWB) comprises 12 items, each on a 0 ('Not at All') to 4 ('Very Much'). The SWB total score is derived by summing the responses, with a higher score representing high spiritual well-being. The minimum score is 0 and the maximum score is 48.
Time Frame: baseline meaning making measures and again at post-intervention (approximately week 8)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Individual Meaning-Centered Psychotherapy (IMCP) | Standard Individual Supportive Psychotherapy (ISP) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 109 | 108 | 104
scores on a scale
  SWB Total Score at Baseline | 28.48 (10.43) | 28.19 (9.31) | 29.53 (8.92)
  SWB Total Score at Post-intervention | 34.59 (9.39) | 32.86 (8.90) | 31.88 (8.28)

3. Secondary Outcome: The Relative Impact of Individual Meaning-Centered Psychotherapy on Different Aspects of Meaning (e.g., Purpose, Coherence, Existential Vacuum), as Well as on Different Aspects of Spiritual Well-being (Meaning Versus Faith),
Description: Single Item Scale (SIS) from the McGill Quality of Life Questionnaire (MQOL): The McGill Quality Of Life Questionnaire is a 17-item scale, with each item rated on a scale of 0 to 10, divided into four domains (the Single-Item Scale (SIS), physical symptoms, feelings and thoughts, and social). It is a brief, self-report instrument designed to assess various domains of psychological, spiritual, and physical functioning among terminally ill patients. In this study the SIS from the MQOL was used. For each scale participants rate their current functioning on a scale of 0 to 10, 0 being Very Bad and 10 being Excellent, higher is better.
Time Frame: baseline meaning making measures and again at post-intervention (approximately week 8)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Individual Meaning-Centered Psychotherapy (IMCP) | Standard Individual Supportive Psychotherapy (ISP) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 109 | 108 | 104
scores on a scale
  MQOL: Physical symptoms at Baseline | 3.73 (2.06) | 3.96 (2.00) | 3.53 (2.18)
  MQOL: Physical symptoms at Post-intervention | 3.76 (2.17) | 3.61 (2.04) | 3.58 (1.96)
  Psychological at Baseline | 6.43 (1.75) | 6.77 (1.71) | 6.78 (1.74)
  Psychological at Post-intervention | 8.08 (1.61) | 7.43 (1.82) | 7.22 (1.63)
  Existential at Baseline | 6.71 (1.75) | 6.77 (1.71) | 6.78 (1.74)
  Existential at Post-intervention | 8.08 (1.61) | 7.43 (1.82) | 7.22 (1.63)
  Overall at Baseline | 6.29 (1.49) | 6.19 (1.55) | 6.24 (1.58)
  Overall at Post-intervention | 7.33 (1.75) | 6.55 (1.59) | 6.49 (1.47)

4. Secondary Outcome: Whether an Enhanced Sense of Meaning "Explains" (Mediates) Improved Psychological Well-being (i.e., Increased Quality of Life, Decreased Psychological Distress).
Description: The Schedule of Attitudes towards Hastened Death (SAHD) comprises 20 TRUE/FALSE questions on the presence or absence of attitudes towards hastened death. A scale score is derived by tallying the number of items endorsed. The minimum score is 0 (better, no thoughts on hastened death) and the maxim score is 20 (worst, many thoughts on hastened death).
Time Frame: 4 years
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Individual Meaning-Centered Psychotherapy (IMCP) | Standard Individual Supportive Psychotherapy (ISP) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 109 | 108 | 104
scores on a scale
  SAHD Total Scores at Baseline | 2.89 (3.16) | 2.95 (3.12) | 2.19 (2.33)
  SAHD Total Scores at Post-intervention | 1.97 (2.26) | 2.62 (2.92) | 2.05 (3.09)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Individual Meaning-Centered Psychotherapy (IMCP) | Standard Individual Supportive Psychotherapy (ISP) | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 9/109 | 15/108 | 5/104
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/108 | 0/104
Other Adverse Events (participants affected / at risk) | 1/109 | 2/108 | 4/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Individual Meaning-Centered Psychotherapy (IMCP) (N=109) | Standard Individual Supportive Psychotherapy (ISP) (N=108) | Enhanced Usual Care (EUC) (N=104)
Distress during assessment (General disorders) | 1 | 2 | 4
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT01323309/Prot_SAP_001.pdf
  • Informed Consent Form (2015-11-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT01323309/ICF_000.pdf